CLINICAL TRIAL: NCT01203137
Title: Prognostic Value of Early Postoperative Right Ventricular Systolic Function in Patients With Isolated Severe Tricuspid Regurgitation
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyung-Kwan Kim, Professor, Seoul National University Hospital
Other Study IDs: H-1009-014-331
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Tricuspid Regurgitation
Keywords: tricuspid regurgitation, severe
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- tricuspid regurgitation, severe: To be included in the present study, the following 3 criteria for severe TR should be met based on the preoperative echocardiography: (1) TR jet > 30% of right atrial area, (2) inadequate cusp coaptation, and (3) systolic flow reversal in the hepatic vein.

SUMMARY:
Preoperative right ventricular end-systolic area (RV-ESA) and hemoglobin level were suggested as independent prognosticator for predicting long-term prognosis in patients with isolated severe TR undergoing corrective surgery We attempted to explore whether early postoperative echocardiography provides additional prognostic information on top of preoperative clinical and echocardiographic variables.

DETAILED DESCRIPTION:
We prospectively recruited patients with isolated severe TR undergoing corrective surgery. Comprehensive preoperative echocardiography was performed in all patients, with the performance of early postoperative echocardiography in all patients. During follow-up, clinical events, defined as operative mortality (death within 30 days after surgery or before discharge), cardiovascular death, repeated open heart surgery, and readmission due to cardiovascular problems were investigated.

ELIGIBILITY:
Inclusion Criteria:

* severe tricuspid regurgitation

Exclusion Criteria:

* concomitant left-sided valve surgery
* significant coronary artery disease

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We prospectively recruited consecutive patients with isolated (without any other valvular dysfunction) severe TR who underwent corrective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
clinical event | 40 months
  Clinical events were defined as operative mortality (death within 30 days after surgery or before discharge), cardiovascular death, repeated open heart surgery, and readmission due to cardiovascular problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea